CLINICAL TRIAL: NCT03146533
Title: Phase I/II Study of CD19 CART Cells for Patients With Relapse and Refractory CD19+ B-cell Lymphoma.
Brief Title: CD19 CART Cells for Patients With Relapse and Refractory CD19+ B-cell Lymphoma.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: The Beijing Pregene Science and Technology Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstShenzhen01
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CART (Experimental): patients will receive a pre-conditioning with cyclophosphamide and fludarabine before infusion of CD19 CART cells. The CD19 CART cells are to be administered on day0,day1,day2.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CD19 CART

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2/day IV for 3 days.
Drug: Cyclophosphamide — patients will receive a standard pre-conditioning regime with cyclophosphamide 0.8g/m2/day IV for 2 days.
Biological: CD19 CART — CD19 CART cells will be administered using a split dose on day0(10%), 1(30%), and 2(60%) after completion of the chemotherapy.

SUMMARY:
This is a clinical study to observe the maximum tolerated dose (MTD) and the safety and feasibility of chimeric antigen receptor 19 (CD19 CART) cells in relapsed and refractory patients with CD19+ B cell lymphoma.

DETAILED DESCRIPTION:
This is a study for the patients with B cell lymphoma. Maximum tolerated dose climbing test is expected into the group of 9 cases of patients. And Phase II expected into the group of 11 subjects, selected the above safe dose, carrying out a research into the clinical effectiveness. Subjects will be collected their T cells and modify them, the modification is a genetic change, that CD19:4-1BB:CD28:CD3 modified T cells, in order to tells the T cells to recognize their target tumor cells and potentially kill them, but not other normal cells in the subject's body. The CART cells will then be expanded in vitro and then administered to subjects. The purpose of this study is observe the MTD and to assess the safety and feasibility of CART cells in the patients with relapsed and refractory CD19+ B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years to 70 years, expected survival > 3 months;
* 2. CD19 positive B-cell lymphoma;
* 3. KPS >80;
* 4. Having at least one measurable lesions;
* 5. Cardiac function: 1-2 levels; Liver: TBIL≤3ULN，AST ≤2.5ULN，ALT ≤2.5ULN; kidney: Cr≤1.25ULN; bone marrow: WBC ≥ 3.0×109/L, Hb ≥90 g/L, PLT ≥ 80×109/L）;
* 6. No serious allergic constitution;
* 7. No other serous diseases that conflicts with the clinical program;
* 8. No other cancer history;
* 9. No serious mental disorder;
* 10. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

* 1. Pregnant or lactating women; (female participants of reproductive potential must have a negative serum or urine pregnancy test);
* 2. Uncontrolled active infection, HIV infection, syphilis serology reaction positive;
* 3. Active hepatitis B or hepatitis C infection;
* 4. Recent or current use of glucocorticoid or other immunosuppressor;
* 5. With severe cardiac, liver, renal insufficiency, diabetes and other diseases;
* 6. Transaminase >2.5ULN, Bilirubin >3ULN，Creatinine>1.25ULN
* 7. Participate in other clinical research in the past three months; previously treatment with any gene therapy products;
* 8. Researchers think of that does not fit to participate in the study, or other cases that affect the clinical trial results;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
safety as assessed by the occurence of study related adverse events | 6 months
  monitor the occurence of study related adverse events
observe the maximum tolerated dose (MTD) | 2 months
objective response rate | 2 years
  CR+PR
disease control rate | 2 years
  CR+PR+SD
overall survival | 2 years
  OS
Progression-Free Survival | 2 years

SECONDARY OUTCOMES:
Determine duration of in vivo survival of CD19 CART cells | 2 years
  CD19 CART vector sequences will be performed by Q-PCR
Peripheral blood cytokines | 2 months
  IL-6、IL-10、IFN-γ、TNF-α
subgroup of T cell | 2 years
  CD3、CD4、CD8

CONTACTS AND LOCATIONS:
Overall Officials: geng tian, Principal Investigator — Shenzhen Second People's Hospital
Locations (1):
- The Second People's Hospital of Shenzhen, Shenzhen, Guangdong, China